CLINICAL TRIAL: NCT03538002
Title: Does Blue-light Filtering Spectacle Lens Promote Myopia Progression in Schoolchildren
Brief Title: The Effect of Blue-light Filtering Spectacle Lenses on Myopia Progression in Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05161146
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-01

CONDITIONS: Myopia
Keywords: blue light filtering spectacle lens
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional anti-reflection coated spectacle lens (No Intervention): Single vision lenses with correction of distant refraction and conventional anti-reflection coating
- Blue-light filtering spectacle lenses (Experimental): Single vision lenses with correction of distant refraction and blue-light filtering coating
  Interventions: Device: Blue-light filtering spectacle lenses

INTERVENTIONS:
Device: Blue-light filtering spectacle lenses — This is a single vision spectacle lens for correction of distant refractions and filtering out the blue light by providing anti-blue light coating.
  Arms: Blue-light filtering spectacle lenses

SUMMARY:
The purpose of this study is to investigate if the blue-light filtering spectacle lenses promote myopia progression in schoolchildren.

DETAILED DESCRIPTION:
The effect of blue light on ocular health has been studied extensively. Shorter wavelength such as blue light could cause damage to the retina. The damage was more evident in the ageing eye. Since the tablets and mobile with blue LED backlight display are widely used, thus blue-light filtering spectacle lenses are now available in the market. However, whether this kind of lenses could affect the eye growth in schoolchildren is unknown. This study is then designed to investigate if the blue-light filtering spectacle lenses affect myopia progression in Hong Kong Chinese schoolchildren. The schoolchildren will be randomly allocated to either blue-light filtering spectacle lens group (treated) or conventional spectacle lens group (control). Their axial length and refraction will be monitored every 6 months for 2 years. The changes between two group will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* Refraction: myopia of -1.00 dioptres (D) to -5.00D
* Astigmatism: equal or less than -1.50D
* Anisometropia: equal or less than 1.00D
* Best corrected monocular visual acuity: 0.0 LogMAR or better after full correction
* Parents' understanding and acceptance of random allocation of grouping

Exclusion Criteria:

* any ocular and systemic abnormalities might affect visual functions or refractive development
* prior treatment of myopic control, e.g. drugs, orthokeratology, progressive addition lenses, bifocal lenses, drugs (e.g. atropine), etc.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Cycloplegic refraction | 2 years
  Refraction done under cycloplegia

SECONDARY OUTCOMES:
Axial length | 2 years
  Length of eyeball that is directly related to myopia

CONTACTS AND LOCATIONS:
Overall Officials: Ka Man Chun, PhD, Principal Investigator — Centre for Myopia Research, The Hong Kong Polytechnic University
Locations (1):
- Centre of Myopia Research, School of Optometry, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No